CLINICAL TRIAL: NCT03966976
Title: Comparison Between "Conventional Monitoring" Versus "Monitoring Via Vitaphone" in the Detection of Post Ablation Atrial Arrhythmias of Paroxysmal Atrial Fibrillation
Acronym: VITAPHONE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: Dr Alexis MECHULAN (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-A01813-50
Record Dates: First submitted 2019-05-28; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitaphone Arm (Experimental): Follow-up via VITAPHONE in addition to conventional monitoring.
  Interventions: Device: ECG monitoring & record
- Conventional Arm (Active Comparator): Conventional follow-up
  Interventions: Other: Conventional follow-up

INTERVENTIONS:
Device: ECG monitoring & record — This is a mobile ECG recorder that not only records short portions of ECG on one or three leads, but also stores, processes and transmits their data to facilitate the diagnosis and to confirm the occurrence of AF arrhythmia episodes by the physician.
  Arms: Vitaphone Arm
Other: Conventional follow-up — Conventional follow-up
  Arms: Conventional Arm

SUMMARY:
Atrial fibrillation (AF) is the most common atrial arrhythmia. Ablation of AF is a recent technique, nevertheless, the success rates of ablation vary between 50% and 70% depending on the paroxysmal or persistent nature of AF. These rates are difficult to assess in routine practice because they are based on the recurrence of fibrillation.

The Vitaphone is a non-invasive device, with which the patient can record a single-track ECG as his or her symptoms take place. The plot is then transmitted via the internet to the centre, which can thus diagnose a relapse of AF.

The aim of our study is to correlate the rhythm and symptoms of 20 patients with Vitaphone 6 months after AF ablation and to compare them with 20 other patients receiving conventional monitoring.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common atrial arrhythmia in the population and its incidence will increase in the coming years. Ablation of AF is a recent technique, the efficiency of which has considerably increased in recent years. Nevertheless, the success rates of ablation vary between 50% and 70% depending on the paroxysmal or persistent nature of AF. These rates are difficult to assess in routine practice because they are based on the recurrence of fibrillation.

This definition of recurrence based on symptoms (palpitations, asthenia, fatigue, shortness of breath, malaise, precordialgia) is widely debated because some patients have asymptomatic AF recidivism, while others experience palpitations that are not due to AF.

In this context, studies have been carried out with electrocardiographic recording devices implanted subcutaneously. Given the invasiveness of this monitoring, it is not feasible in current practice.

The Vitaphone is a non-invasive device, with which the patient can record a single-track ECG as his or her symptoms take place. The plot is then transmitted via the internet to the centre, which can thus diagnose a relapse of AF.

The aim of our study is to correlate the rhythm and symptoms of 20 patients with Vitaphone 6 months after AF ablation and to compare them with 20 other patients receiving conventional monitoring.

This is, to our knowledge, the first non-invasive French study using the Vitaphone.

ELIGIBILITY:
Inclusion Criteria:

* AF ablated patient
* Patient with paroxysmal AF before the procedure
* Patient with health insurance or beneficiary of a social security scheme
* Unprotected adult patient
* Patient having given their consent

Exclusion Criteria:

* Patient having undergone an AF ablation due to persistent AF
* Unable to understand or handle the Vitaphone alone
* Failure to participate
* Minors
* Pregnant, lactating or parturient women
* Adult receiving psychiatric care, under legal protection, trusteeship or guardianship, or deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of AF between 3 and 6 months | 3 to 6 months
  Atrial arrhythmia documented in each arm by either an ECG or Holter or Vitaphone between 3 and 6 months post-ablation of paroxysmal AF and validated by a cardiologist.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis MECHULAN, Principal Investigator — CRRIC Clairval Hospital
Locations (1):
- CRRIC Clairval Interventional Rhythmology Research Centre Clairval Private Hospital, Marseille, PACA, France

IPD SHARING:
Plan to Share IPD: No